CLINICAL TRIAL: NCT04188210
Title: Elbow Pain in Hemodialysis Patients and Its Effect on Daily Living Activities of the Patients
Status: Completed | Type: Observational
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Betül Tepeli, Department of Physical Medicine And Rehabilitation, Private Balkan Hospital,Principal Investigator,, Namik Kemal University
Other Study IDs: 2019
Record Dates: First submitted 2019-11-29; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: End Stage Renal Disease
Keywords: musculoskeletal pain; elbow pain; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Presence of elbow pain in patients with end stage renal disease — The Beck Depression Inventory (BDI), the Nottingham Health Profile (NHP) scores were measured for all patients to evaluate depression symptoms and health-related quality of life. The elbow pain presence was asked to all the patients, the patients with elbow pain were also evaluated with The Disabilities of the Arm, Shoulder and Hand Score (Q-DASH) and Visual Analogue Scale (VAS). VAS detected as pain during rest, activity, night and pain at last week.

SUMMARY:
The study will include the patients undergoing hemodialysis.

DETAILED DESCRIPTION:
The study will include the patients undergoing hemodialysis. The patients with surgery at upper extremity in last 3 months, the presence of conditions such as cancer, chronic hearing loss and neurologic diseases affect the interview will be excluded. Sociodemographic properties which include age, gender, duration of dialysis, educational level, comorbid diseases, vascular access area, hand dominancy will be asked. The Beck Depression Inventory (BDI), the Nottingham Health Profile (NHP), the Disabilities of the Arm, Shoulder and Hand Score (Q-DASH) and Visual Analogue Scale (VAS) will applied to all patients.

All the demographic results and vascular access area for hemodialysis will be detected. All data for normality will be tested by using Kolmogorov-Smirnov test. To compare the differences between groups, Mann Whitney U test will be used

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old having hemodialysis treatment

Exclusion Criteria:

* any surgical operation at upper extremity in last 3 months, the presence of conditions such as cancer, chronic hearing loss and neurologic diseases can affect the interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with end stage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Kolmogorov-Smirnov test | through study completion, an average of 1 month
  All data for normality was tested by using Kolmogorov-Smirnov test

CONTACTS AND LOCATIONS:
Overall Officials: betül tepeli, Principal Investigator — private balkan hospital
Locations (1):
- Private Balkan Hospital, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fidan F, Alkan BM, Tosun A, Altunoglu A, Ardicoglu O. Quality of life and correlation with musculoskeletal problems, hand disability and depression in patients with hemodialysis. Int J Rheum Dis. 2016 Feb;19(2):159-66. doi: 10.1111/1756-185X.12171. Epub 2013 Oct 31. PMID 24176031
- [Result] Kane SF, Lynch JH, Taylor JC. Evaluation of elbow pain in adults. Am Fam Physician. 2014 Apr 15;89(8):649-57. PMID 24784124